CLINICAL TRIAL: NCT05196763
Title: Maximizing the Impact of Nutrition Education to Meet the Dietary Quality and Food Security Needs of Children and Parents
Brief Title: Maximizing Nutrition Education to Meet Dietary and Food Security of Children and Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Heather Eicher-Miller, Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIFA 2022-68015-36279
Record Dates: First submitted 2021-12-16; First posted 2022-01-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Nutrition, Healthy; Hunger; Diet, Healthy; Food Habits
Keywords: food security; food insecurity; dietary quality; nutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: 2-arm, intervention and control, parallel design, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplemental Nutrition Assistance Program-Education (Experimental): This group will receive the core content of the Supplemental Nutrition Assistance Program-Education over the 10-week "intervention period".
  Interventions: Behavioral: the Supplemental Nutrition Assistance Program-Education
- Control (No Intervention): This group will not receive the Supplemental Nutrition Assistance Program-Education during the "intervention period" nor throughout the study (1 year).

INTERVENTIONS:
Behavioral: the Supplemental Nutrition Assistance Program-Education — The Supplemental Nutrition Assistance Program-Education is federal nutrition education provided in all U.S. states to the SNAP-eligible population.
  Arms: Supplemental Nutrition Assistance Program-Education

SUMMARY:
Food insecurity and low diet quality are persistent problems linked with chronic disease and poor health among limited-resource children and adults using Supplemental Nutrition Assistance Program (SNAP). We have shown nutrition education via adult-focused, direct SNAP-Education (SNAP-Ed) improved household food security by 25% but not adult dietary quality among SNAP-eligible households using a randomized, controlled, longitudinal SNAP-Ed intervention in Indiana. Households experiencing food insecurity often reserve food considered "healthful" for children, so child dietary quality improvement may precede that observed among adults when household food security improves. This study will determine the effect of adult-focused direct SNAP-Ed on child dietary quality and household food security using a longitudinal randomized, controlled SNAP-Ed intervention. Assessment will include repeated 24-hour dietary recalls to determine usual intake, the U.S. Household Food Security Survey Module, and behavior data from before and after the 10-week "intervention period," and 1 year later, after which the control group will receive the intervention. Low-income participants (n=275) from Indiana will be recruited following SNAP-Ed protocol. Results of the study will inform the creation of supplementary on-demand SNAP-Ed educational material focused on improving healthful dietary intake for children and adults in situations of food insecurity in households with children. Education on modeling healthy attitudes and behaviors, planning and preparing family meals, and dietary shortfalls as informed by the results and previous evidence will be included and evaluated. The study aligns with the goals of USDA to increase food security and this RFP to improve healthful behaviors, food quality and nutrition.

DETAILED DESCRIPTION:
The goals of SNAP-Ed are to "improve the likelihood that persons eligible for SNAP will make healthy choices… consistent with the current Dietary Guidelines for Americans." Our recent review found four studies evaluating household food security as an outcome of direct adult SNAP-Ed with evidence considered strong because of our studies that used randomized and controlled study designs and assessment using the U.S. Household Food Security Survey Module (HFSSM).We showed that nutrition education via adult-focused, direct SNAP-Ed improved household food security by 25% among SNAP-eligible households over 1 year after a SNAP-Ed intervention in Indiana. However, previous evidence of meaningful change in dietary quality and intake among adult SNAP-Ed recipients is less secure despite demonstrated changes in attitudes, self-efficacy, intentions, and behaviors toward increasing intake of nutrient-dense foods due to a lack of randomized, controlled, longitudinal study designs and inherent measurement error in the assessments quantifying diet. Importantly, our study, using a longitudinal, randomized, controlled design and estimating usual intake with best practice assessment and analysis, did not determine dietary quality change among adults nor other dietary components except for vitamin D. Households experiencing food insecurity often reserve food considered "healthful" for children so child dietary quality improvement may proceed that observed among adults when household food security is improved. As children age, however, diets are known to worsen. Therefore, dietary quality improvement over time due to SNAP-Ed will need to overcome a strong influence of age, yet even maintained dietary quality over time would be a success compared to the expected declines in dietary quality for a control group whose parents do not receive SNAP-Ed. Taken together, we hypothesize that dietary quality among children and household food security will improve 1 year after a direct, adult-focused SNAP-Ed intervention compared with a control group while adult dietary quality will not improve compared with the control group.

Long-Term Goal: Determine the long-term (1-year) effect of direct, adult-focused SNAP-Ed on dietary quality and household food security among children (5-18 years) of adult (≥18 years), low-income Indiana SNAP-Ed participants.

(a) dietary quality (using the HEI), usual dietary intake, among children of adult SNAP-Ed participants and the adult participants themselves, compared with a control group receiving a delayed intervention and (b) food security among the household, adults and children (using the U.S. HFSSM) in intervention compared with control group, and (c) coping mechanisms, needs, behaviors, and attitudes among adult SNAP-Ed participants compared with controls.

1. Objectives Research Objectives

1. Recruit and randomize n=275 SNAP qualifying, low-income adult (≥18 years) and child (5-18 years) pairs from Indiana to participate in this longitudinal study with approximately n=138 pairs receiving the SNAP-Ed intervention and n=138 pairs in the control group (not receiving SNAP-Ed until after the study).
2. Quantify child and adult dietary quality (HEI) and usual intake (2, 24-hour recalls at each time-point), household, adult and child food security, and additional behavioral, coping mechanisms, needs, and self-efficacy at baseline and 1 year after the intervention period.
3. Evaluate change in child and adult dietary quality and usual intake per DGA compliance and food components of public health relevance (as per Dietary Reference Intake standards); household, adult and child food security status; from baseline one year follow-up for intervention compared with control group. Due to nonresponse and loss-to-follow, we expect roughly 100 pairs in each group to provide change measures.

Goal 1:Research Study Participants and Recruitment Recruitment will occur at a rate of n=10 per week for 9 months in the 4 regions of the state (northwest, northeast, southwest, southeast) over the course of the school year so that each region is visited roughly once per month to avoid a seasonal effect. Approved SNAP-Ed sites within regions will serve as recruitment sites including community centers; SNAP, WIC, county Extension offices; food pantries and banks, and other locations. An informational flyer will be posted at the site on study recruitment days. A full-time study recruiter, trained through SNAP-Ed, will coordinate to recruit alongside the NEPAs in the 4 state regions who will be present to similarly recruit for SNAP-Ed programming and deliver the lessons. The recruiter will explain the study procedures, assessments, and time necessary to complete the assessments. The recruiter will gauge interest and administer the screener querying exclusion criteria. The consent form, randomization, and study assessments will follow if the individual desires to participate, if not they will be referred to the NEPA and engage in SNAP-Ed as usual without differential treatment through the program. Assent for children 5-17 years and consent for children 18 years and assessments will be scheduled with the recruiter within the following 24 hours by phone or by email when the participant desires. Participants joining the study will be queried as to whether they prefer assessment via interview or independently online and similarly their preference for completing the 1-year assessments. The reason for any non-response will be tracked if known. Participants without email, without access to a computer with internet, or with limited computer skills may also complete the assessments via telephone with assistance from researchers. Treatment group (control or SNAP-Ed intervention) will be assigned 1:1 using data collection spreadsheets that will include the subject ID and randomized assignment. Participants recruited simultaneously will be assigned to the same study group to prevent knowledge of differential treatment. Subject ID will be assigned to each assessment the participant completes; names will not be associated with any assessments, and the list of names and numbers will be kept separately and securely. A password protected metadata file on an encrypted hard drive or REDCap or Box will securely store all information.

Research Study Protocols: Adult participants will complete assessments following recruitment. The participant screener, characteristics and additional behavioral, coping mechanisms, needs, self-efficacy, and food security questionnaires will be completed online or interview assisted in Qualtrics or REDCap. Child participants will complete the child-specific questions of the U.S. HFSSM, and a brief set of behavioral, and coping mechanisms questionnaires online (with interview and parent assistance for ages 6-11 years and with interview and option to self-complete for ages 12-18 years). Study assessments for the intervention group will be provided alongside the SNAP-Ed program evaluation before the first lesson. The 24-hour dietary recall will be self-completed online or via interview for adults using the Automated Self-Administered 24-hour (ASA-24) Dietary Recall and by interview with parent assistance ages 6-11 years and by interview or self-completed for ages 12-18 years through a secure data management system. The same sequence of assessments will be completed at each time point, with the exception of the participant screener completed at baseline. Assessments will include: (1) participant screener, characteristics, behavioral, coping mechanisms, needs, self-efficacy, and U.S. HFSSM using a 1-year reference period and (2) SNAP-Ed curricula program evaluation, (3) recruitment day dietary assessment using a 24-hour dietary recall for adult and child, and (4) non-consecutive day follow-up dietary recall for adult and child. The characteristics portion of the survey will query personal and household characteristics.

After baseline study assessments are completed, participants randomized and recruited to the intervention group will be referred to the SNAP-Ed NEPA and receive the first SNAP-Ed lesson. The remaining 3 lessons will be received at the rate of 1 lesson per week during the 10 week intervention period, following normal protocol. Control group participants will not receive lessons during the intervention period and will be requested to wait 1 year to receive lessons. All recruited participants (control and intervention groups) will be contacted at least once per month via communication of their choice to reduce attrition and maintain correct contact information until completion of the final survey. SNAP-Ed lessons will be delivered either one-on-one or in a group setting at a community location, following normal protocol.

The study recruiter will follow-up with NEPAs delivering lessons to intervention participants to track lesson attendance, location, NEPA delivering the lessons, delivery to individual or group, contacts with the NEPA, and presence and type of county-level indirect SNAP-Ed for each participant using a spreadsheet in Qualtrics or RedCAP. Next, the study recruiter will request to keep in touch with each participant to update contact information on a monthly basis to minimize attrition. After 1-year, participants will complete 1-year assessments and the control-group referred to SNAP-Ed.

Success of the randomization for the Goal 1 will be checked by comparison of the experimental group with the control group for each measured independent variable for all characteristics variables and potential confounders. The interaction of time and treatment group in this model will be the main independent variable of interest while the various outcomes will be the main dependent variables in different models. The difference of differences will be determined by comparing changes in outcomes from baseline to the 1-year follow-up in each treatment group using linear contrasts. The model conditions necessary for inference will be checked through residual plots, Q-Q plots, and histograms. Remedial measures such as transformations, will be completed to address non-normal distributions. Least squares mean estimates of the 1-year change by treatment group and their difference (i.e., the interaction) will be reported along with their standard errors. Results will be significant when p≤0.05 performed using SAS.

Dietary quality and intake: Adult and child participants with at least one complete ASA-24 recall and complete baseline survey information will be included in the analysis of diet quality and intake. Outcomes will be the difference of the change in usual dietary quality and component scores and usual intakes by time between the intervention and the control group for nutrients and food groups of interest, and the proportions of the study group not meeting the DGA, EAR, or exceeding the AI. To assess overall diet quality, the HEI-2015 scores will be analyzed between groups over time. The NCI method will be used to estimate distributions of usual intakes and the proportion of the population at risk for nutrient inadequacy based on the cut-point method and probability method for iron. Models will be adjusted for covariates treated as fixed effects: age, energy as kilocalories, and variables indicating the day of the week of the recall (weekday (Monday-Thursday) or weekend day (Friday-Sunday)) and the sequence of the recall (1st or 2nd). Other covariates described for food security models will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* households in Indiana
* households with children
* English speaking
* eligible to receive SNAP (≥18 years and household income at or below 130% of the poverty guideline)
* willing to allow a child 5-18 years to participate
* willing to participate in the study and wait 1 year to receive SNAP-Ed

Exclusion Criteria:

* not have received SNAP-Ed lessons in the past year
* not pregnant or lactating (due to inherent dietary changes)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in food security from baseline to 12 months | food security of the previous 12 months at baseline and 12 months later
  Determined based on the 18-item US Household Food Security Survey Module
Change in dietary quality from baseline to 12 months | Two 24-hour dietary recalls on two non-consecutive days at baseline and 12 months later
  Determined based on the Healthy Index Score, where 100 indicates complete alignment with the Dietary Guidelines for Americans and 0 is the minimum score, as calculated from two 24-hour dietary recalls
Change in usual dietary intake of food groups and nutrients | Two 24-hour dietary recalls on two non-consecutive days at baseline and 12 months later
  Determined based on two, 24-hour dietary recalls asking about intake of all foods and beverages consumed

CONTACTS AND LOCATIONS:
Overall Officials: Heather Eicher-Miller, PhD, Principal Investigator — Purdue University
Locations (1):
- Heather Eicher-Miller, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conrad Z, Rehm CD, Wilde P, Mozaffarian D. Cardiometabolic Mortality by Supplemental Nutrition Assistance Program Participation and Eligibility in the United States. Am J Public Health. 2017 Mar;107(3):466-474. doi: 10.2105/AJPH.2016.303608. Epub 2017 Jan 19. PMID 28103061
- [Background] Nguyen BT, Shuval K, Bertmann F, Yaroch AL. The Supplemental Nutrition Assistance Program, Food Insecurity, Dietary Quality, and Obesity Among U.S. Adults. Am J Public Health. 2015 Jul;105(7):1453-9. doi: 10.2105/AJPH.2015.302580. Epub 2015 May 14. PMID 25973830
- [Background] Singh GK, Miller BA, Hankey BF, Edwards BK. Area socioeconomic variations in US cancer incidence, mortality, stage, treatment, and survival, 1975-1999. NCI Cancer Surveillance Monograph Series, Number 4. Bethesda, MD: National Cancer Institute, 2003. NIH Publication No. 03-5417.
- [Background] U.S.Department of Agriculture and U.S. Department of Helth and Human Services. Dietary Guidelines for Americans 2020-2025. 9th Edition. December 2020. Available at: https://www.dietaryguidelines.gov/sites/default/files/2020-12/Dietary_Guidelines_for_Americans_2020-2025.pdf (Accessed on 23 May 2021)
- [Background] Dietary Guidelines Advisory Committee. 2020. Scientific Report of the 2020 Dietary Guidelines Advisory Committee: Advisory Report to the Secretary of Agriculture and the Secretary of Health and Human Services. U.S. Department of Agriculture, Agricultural Research Service, Washington, DC. Available at: https://www.dietaryguidelines.gov/2020-advisory-committee-report (Accessed on 23 May 2021)
- [Background] Reedy J, Lerman JL, Krebs-Smith SM, Kirkpatrick SI, Pannucci TE, Wilson MM, Subar AF, Kahle LL, Tooze JA. Evaluation of the Healthy Eating Index-2015. J Acad Nutr Diet. 2018 Sep;118(9):1622-1633. doi: 10.1016/j.jand.2018.05.019. PMID 30146073
- [Background] Nguyen BT, Shuval K, Njike VY, Katz DL. The Supplemental Nutrition Assistance Program and dietary quality among US adults: findings from a nationally representative survey. Mayo Clin Proc. 2014 Sep;89(9):1211-9. doi: 10.1016/j.mayocp.2014.05.010. Epub 2014 Aug 5. PMID 25107469
- [Background] Coleman-Jensen A, Rabbitt MP, Gregory CA, and Singh A. 2020. Household food security in the United States in 2019, ERR-275, U.S. Department of Agriculture, Economic Research Service. Available at: https://www.ers.usda.gov/webdocs/publications/99282/err-275.pdf?v=7113.8 (Accessed on 23 May 2021).
- [Background] Core indicators of nutritional state for difficult-to-sample populations. J Nutr. 1990 Nov;120 Suppl 11:1559-600. doi: 10.1093/jn/120.suppl_11.1555. PMID 2243305
- [Background] Hanson KL, Connor LM. Food insecurity and dietary quality in US adults and children: a systematic review. Am J Clin Nutr. 2014 Aug;100(2):684-92. doi: 10.3945/ajcn.114.084525. Epub 2014 Jun 18. PMID 24944059
- [Background] Gundersen C, Ziliak JP. Food Insecurity And Health Outcomes. Health Aff (Millwood). 2015 Nov;34(11):1830-9. doi: 10.1377/hlthaff.2015.0645. PMID 26526240
- [Background] Cook J, Poblacion AP. Estimating the health-related costs of food insecurity and hunger. Bread for the World Institute. 2016. Available at: http://hungerreport.org/costofhunger/ (Accessed on 23 May 2021).
- [Background] Feeding America. The impact of the coronavirus pandemic on food insecurity in 2020 & 2021. March 2021. Available at: https://www.feedingamerica.org/sites/default/files/2021-03/National%20Projections%20Brief_3.9.2021_0.pdf (Accessed on 23 May 2021).
- [Background] Rajgopal R, Cox RH, Lambur M, Lewis EC. Cost-benefit analysis indicates the positive economic benefits of the Expanded Food and Nutrition Education Program related to chronic disease prevention. J Nutr Educ Behav. 2002 Jan-Feb;34(1):26-37. doi: 10.1016/s1499-4046(06)60225-x. PMID 11917669
- [Background] United States Department of Agriculture, National Institute of Food and Agriculture. Supplemental Nutrition Education Program-Education (SNAP-Ed). Available at: https://nifa.usda.gov/program/supplemental-nutrition-education-program-education-snap-ed. (Accessed on 23 May 2021).
- [Background] Lambur MT, Rajgopal R, Lewis EC, Cox RH, Ellerbrock M. Applying cost benefit analysis to nutrition education programs: Focus on the Virginia Expanded Food and Nutrition Education Program. 1999. Available at: https://vtechworks.lib.vt.edu/bitstream/handle/10919/50174/490-403.pdf? sequence=1. (Accessed on 21 May 2021).
- [Background] Dollahite J, Kenkel D, Thompson CS. An economic evaluation of the expanded food and nutrition education program. J Nutr Educ Behav. 2008 May-Jun;40(3):134-43. doi: 10.1016/j.jneb.2007.08.011. PMID 18457781
- [Background] Rivera RL, Maulding MK, Abbott AR, Craig BA, Eicher-Miller HA. SNAP-Ed (Supplemental Nutrition Assistance Program-Education) Increases Long-Term Food Security among Indiana Households with Children in a Randomized Controlled Study. J Nutr. 2016 Nov;146(11):2375-2382. doi: 10.3945/jn.116.231373. Epub 2016 Sep 28. PMID 27683869
- [Background] Rivera RL, Maulding MK, Eicher-Miller HA. Effect of Supplemental Nutrition Assistance Program-Education (SNAP-Ed) on food security and dietary outcomes. Nutr Rev. 2019 Dec 1;77(12):903-921. doi: 10.1093/nutrit/nuz013. PMID 31077323
- [Background] Eicher-Miller HA, Mason AC, Abbott AR, McCabe GP, Boushey CJ. The effect of Food Stamp Nutrition Education on the food insecurity of low-income women participants. J Nutr Educ Behav. 2009 May-Jun;41(3):161-8. doi: 10.1016/j.jneb.2008.06.004. PMID 19411049
- [Background] Kaiser L, Chaidez V, Algert S, Horowitz M, Martin A, Mendoza C, Neelon M, Ginsburg DC. Food Resource Management Education With SNAP Participation Improves Food Security. J Nutr Educ Behav. 2015 Jul-Aug;47(4):374-8.e1. doi: 10.1016/j.jneb.2015.01.012. Epub 2015 Apr 3. PMID 25843204
- [Background] Adedokun OA, Plonski P, Jenkins-Howard B, Cotterill DB, Vail A. Healthy Choices for Every Body Adult Curriculum Improves Participants' Food Resource Management Skills and Food Safety Practices. J Nutr Educ Behav. 2018 Jun;50(6):638-644. doi: 10.1016/j.jneb.2018.02.005. Epub 2018 Apr 3. PMID 29625915
- [Background] Bickel G, Nord M, Price C, Hamilton W, Cook J. Guide to measuring household food security, revised 2000. Alexandria, VA: United States Department of Agriculture, Food and Nutrition Service; 2000.
- [Background] United States Department of Agriculture, Economic Research Service. Survey Tools. Available at: https://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-us/survey-tools/#household (Accessed on 23 May 2021).
- [Background] Qin Y, Rivera RL, Zhang Y, Wang Q, Tooze JA, Abbott AR, Maulding MK, Craig BA, Bailey RL, Eicher-Miller HA. A Randomized Intervention of Supplemental Nutrition Assistance Program-Education Did Not Improve Dietary Outcomes Except for Vitamin D Among Lower-Income Women in Indiana. J Acad Nutr Diet. 2023 Feb;123(2):284-298.e2. doi: 10.1016/j.jand.2022.06.030. Epub 2022 Jun 30. PMID 35781080
- [Background] Radimer KL, Olson CM, Greene J, Campbell CC, Habicht JP. understanding hunger and developing indicators to assess it in women and children. J Nutr Educ. 1992;24 Suppl 1:S36-44.
- [Background] McIntyre L, Glanville NT, Raine KD, Dayle JB, Anderson B, Battaglia N. Do low-income lone mothers compromise their nutrition to feed their children? CMAJ. 2003 Mar 18;168(6):686-91. PMID 12642423
- [Background] Eicher-Miller HA, Park CY, Bailey R. Identifying nutritional gaps among Americans. In: Dietary Supplements in Health Promotion. 2015. 17-54 [TC Wallace, Ed]. Boca Raton, FL: CRN Press.
- [Background] U.S. Department of Agriculture. SNAP-Ed Toolkit. Available at: https://snapedtoolkit.org/ (Accessed on 23 May 2021).
- [Background] Yee AZ, Lwin MO, Ho SS. The influence of parental practices on child promotive and preventive food consumption behaviors: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2017 Apr 11;14(1):47. doi: 10.1186/s12966-017-0501-3. PMID 28399881
- [Background] Romanos-Nanclares A, Zazpe I, Santiago S, Marin L, Rico-Campa A, Martin-Calvo N. Influence of Parental Healthy-Eating Attitudes and Nutritional Knowledge on Nutritional Adequacy and Diet Quality among Preschoolers: The SENDO Project. Nutrients. 2018 Dec 3;10(12):1875. doi: 10.3390/nu10121875. PMID 30513857
- [Background] Dickens E, Ogden J. The role of parental control and modelling in predicting a child's diet and relationship with food after they leave home. A prospective study. Appetite. 2014 May;76:23-9. doi: 10.1016/j.appet.2014.01.013. Epub 2014 Jan 27. PMID 24480669
- [Background] Palfreyman Z, Haycraft E, Meyer C. Development of the Parental Modelling of Eating Behaviours Scale (PARM): links with food intake among children and their mothers. Matern Child Nutr. 2014 Oct;10(4):617-29. doi: 10.1111/j.1740-8709.2012.00438.x. Epub 2012 Aug 20. PMID 22906242
- [Background] Natale RA, Messiah SE, Asfour L, Uhlhorn SB, Delamater A, Arheart KL. Role modeling as an early childhood obesity prevention strategy: effect of parents and teachers on preschool children's healthy lifestyle habits. J Dev Behav Pediatr. 2014 Jul-Aug;35(6):378-87. doi: 10.1097/DBP.0000000000000074. PMID 25007060
- [Background] U.S.Department of Agriculture. Dietary Guidelines for Americans 2015-2020. Available at: https://health.gov/our-work/food-nutrition/2015-2020-dietary-guidelines/guidelines/_(Accessed on 23 May 2021).
- [Background] Indiana Family Nutrition Program Fiscal Year 2019-2020 Report. 2020. Purdue University Health and Human Sciences Extension.
- [Background] Rivera RL, Zhang Y, Wang Q, Maulding MK, Tooze JA, Wright BN, Craig BA, Bailey RL, Eicher-Miller HA. Diet Quality and Associations with Food Security among Women Eligible for Indiana Supplemental Nutrition Assistance Program-Education. J Nutr. 2020 Aug 1;150(8):2191-2198. doi: 10.1093/jn/nxaa171. PMID 32559278
- [Background] Eicher-Miller HA, Rivera RL, Sun H, Zhang Y, Maulding MK, Abbott AR. Supplemental Nutrition Assistance Program-Education Improves Food Security Independent of Food Assistance and Program Characteristics. Nutrients. 2020 Aug 29;12(9):2636. doi: 10.3390/nu12092636. PMID 32872411
- [Background] Rivera RL, Dunne J, Maulding MK, Wang Q, Savaiano DA, Nickols-Richardson SM, Eicher-Miller HA. Exploring the association of urban or rural county status and environmental, nutrition- and lifestyle-related resources with the efficacy of SNAP-Ed (Supplemental Nutrition Assistance Program-Education) to improve food security. Public Health Nutr. 2018 Apr;21(5):957-966. doi: 10.1017/S1368980017003391. Epub 2017 Dec 4. PMID 29199629
- [Background] Neuenschwander LM, Abbott A, Mobley AR. Assessment of low-income adults' access to technology: implications for nutrition education. J Nutr Educ Behav. 2012 Jan-Feb;44(1):60-5. doi: 10.1016/j.jneb.2011.01.004. Epub 2011 Sep 16. PMID 21924959
- [Background] Tooze JA, Kipnis V, Buckman DW, Carroll RJ, Freedman LS, Guenther PM, Krebs-Smith SM, Subar AF, Dodd KW. A mixed-effects model approach for estimating the distribution of usual intake of nutrients: the NCI method. Stat Med. 2010 Nov 30;29(27):2857-68. doi: 10.1002/sim.4063. PMID 20862656
- [Background] Tooze JA, Midthune D, Dodd KW, Freedman LS, Krebs-Smith SM, Subar AF, Guenther PM, Carroll RJ, Kipnis V. A new statistical method for estimating the usual intake of episodically consumed foods with application to their distribution. J Am Diet Assoc. 2006 Oct;106(10):1575-87. doi: 10.1016/j.jada.2006.07.003. PMID 17000190
- [Background] Zhang S, Midthune D, Guenther PM, Krebs-Smith SM, Kipnis V, Dodd KW, Buckman DW, Tooze JA, Freedman L, Carroll RJ. A NEW MULTIVARIATE MEASUREMENT ERROR MODEL WITH ZERO-INFLATED DIETARY DATA, AND ITS APPLICATION TO DIETARY ASSESSMENT. Ann Appl Stat. 2011 Jun 1;5(2B):1456-1487. doi: 10.1214/10-AOAS446. PMID 21804910
- [Background] Kirkpatrick SI, Reedy J, Krebs-Smith SM, Pannucci TE, Subar AF, Wilson MM, Lerman JL, Tooze JA. Applications of the Healthy Eating Index for Surveillance, Epidemiology, and Intervention Research: Considerations and Caveats. J Acad Nutr Diet. 2018 Sep;118(9):1603-1621. doi: 10.1016/j.jand.2018.05.020. PMID 30146072
- [Background] Liu Y, Tooze JA, Zhang Y, Leidy HJ, Bailey RL, Wright B, Ma M, Stluka S, Remley DT, McCormack LA, Franzen-Castle L, Henne R, Mehrle D, Eicher-Miller HA. Breakfast Consumption Is Positively Associated with Usual Nutrient Intakes among Food Pantry Clients Living in Rural Communities. J Nutr. 2020 Mar 1;150(3):546-553. doi: 10.1093/jn/nxz258. PMID 31711170
- [Background] Wright BN, Tooze JA, Bailey RL, Liu Y, Rivera RL, McCormack L, Stluka S, Franzen-Castle L, Henne B, Mehrle D, Remley D, Eicher-Miller HA. Dietary Quality and Usual Intake of Underconsumed Nutrients and Related Food Groups Differ by Food Security Status for Rural, Midwestern Food Pantry Clients. J Acad Nutr Diet. 2020 Sep;120(9):1457-1468. doi: 10.1016/j.jand.2020.04.011. Epub 2020 Jul 20. PMID 32703690
- [Background] Jun S, Thuppal SV, Maulding MK, Eicher-Miller HA, Savaiano DA, Bailey RL. Poor Dietary Guidelines Compliance among Low-Income Women Eligible for Supplemental Nutrition Assistance Program-Education (SNAP-Ed). Nutrients. 2018 Mar 8;10(3):327. doi: 10.3390/nu10030327. PMID 29518042
- [Background] Eicher-Miller HA, Zhao Y. Evidence for the age-specific relationship of food insecurity and key dietary outcomes among US children and adolescents. Nutr Res Rev. 2018 Jun;31(1):98-113. doi: 10.1017/S0954422417000245. Epub 2018 Jan 10. PMID 29318982
- [Background] Campbell CC. Food insecurity: a nutritional outcome or a predictor variable? J Nutr. 1991 Mar;121(3):408-15. doi: 10.1093/jn/121.3.408. PMID 2002411
- [Background] Leung CW, Blumenthal SJ, Hoffnagle EE, Jensen HH, Foerster SB, Nestle M, Cheung LW, Mozaffarian D, Willett WC. Associations of food stamp participation with dietary quality and obesity in children. Pediatrics. 2013 Mar;131(3):463-72. doi: 10.1542/peds.2012-0889. Epub 2013 Feb 25. PMID 23439902
- [Background] United States Department of Agriculture, Food and Nutrition Service. Supplemental Nutrition Assistance Program Education Plan Guidance FY 2022: Nutrition Education and Obesity Prevention Program. 2022. Available at: https://snaped.fns.usda.gov/sites/default/files/documents/FY%202022%20SNAP-Ed%20Plan%20Guidance.pdf . (Accessed on 23 May 2021).
- [Background] Cates S, Blitstein J, Hersey J, Kosa K, Flicker L, Morgan K, Bell L. Addressing the challenges of conducting effective Supplemental Nutrition Assistance Program Education (SNAP-Ed) Evaluations: A step-by-step guide. Prepared by Altarum Institute and RTI International for the U.S. Department of Agriculture, Food and Nutrition Service, March 2014. Available at: https://fns-prod.azureedge.net/sites/default/files/SNAPEDWaveII_Guide.pdf (Accessed on 23 May 2021).
- [Background] United States Department of Agriculture, National Institute of Food and Agriculture SNAP-Ed Budget Allocation, FY 2020. Available at: https://snaped.fns.usda.gov/sites/default/files/documents/FY%202020%20Allocations%20FINAL%2010_08_2019.pdf (Accessed 23 May 2021)
- [Background] Naja-Riese A, Keller KJM, Bruno P, Foerster SB, Puma J, Whetstone L, MkNelly B, Cullinen K, Jacobs L, Sugerman S. The SNAP-Ed Evaluation Framework: demonstrating the impact of a national framework for obesity prevention in low-income populations. Transl Behav Med. 2019 Oct 1;9(5):970-979. doi: 10.1093/tbm/ibz115. PMID 31570929
- [Background] Palmer SM, Knoblauch ST, Winham DM, Hiller MB, Shelley MC. Putting Knowledge into Practice: Low-Income Women Talk about Food Choice Decisions. Int J Environ Res Public Health. 2020 Jul 15;17(14):5092. doi: 10.3390/ijerph17145092. PMID 32679700
- [Background] Fram MS, Frongillo EA, Jones SJ, Williams RC, Burke MP, DeLoach KP, Blake CE. Children are aware of food insecurity and take responsibility for managing food resources. J Nutr. 2011 Jun;141(6):1114-9. doi: 10.3945/jn.110.135988. Epub 2011 Apr 27. PMID 21525257
- [Background] Kamdar N, Rozmus CL, Grimes DE, Meininger JC. Ethnic/Racial Comparisons in Strategies Parents Use to Cope with Food Insecurity: A Systematic Review of Published Research. J Immigr Minor Health. 2019 Feb;21(1):175-188. doi: 10.1007/s10903-018-0720-y. PMID 29549476
- [Background] Rose D, Oliveira V. Nutrient intakes of individuals from food-insufficient households in the United States. Am J Public Health. 1997 Dec;87(12):1956-61. doi: 10.2105/ajph.87.12.1956. PMID 9431283
- [Background] NC Division of Public Health: Nutrition Services Branch and Community and Clinical Connections for Prevention and Health Branch; NC State Extension, NC State University. Families eating smart and moving more (FESMM). Available at: https://ncefnep.org/partners/curricula/ (Accessed on 23 May 2021).
- [Background] U.S. Department of Agriculture, Regional Nutrition Education Centers of Excellence, National Coordination Center at the University of Kentucky. SNAP-Ed Toolkit: Families Eating Smart and Moving More (FESMM). Available at: https://snapedtoolkit.org/interventions/programs/families-eating-smart-and-moving-more-fesmm/ . (Accessed on 23 May 2021).
- [Background] Gregson J, Foerster SB, Orr R, Jones L, Benedict J, Clarke B, Hersey J, Lewis J, Zotz AK. System, environmental, and policy changes: using the social-ecological model as a framework for evaluating nutrition education and social marketing programs with low-income audiences. J Nutr Educ. 2001;33 Suppl 1:S4-15. doi: 10.1016/s1499-4046(06)60065-1. PMID 12857540
- [Background] Bandura A. Social foundations of thought and action. A social cognitive theory. Englewood Cliffs, NJ: Prentice-Hall, 1986.
- [Background] U.S. Department of Agriculture, SNAP-Ed Connection. SNAP Education (SNAP-Ed). Available at: https://snaped.fns.usda.gov/ (Accessed on 23 May 2021).
- [Background] Ajzen I. The theory of planned behavior. Organ Behav Hum Decis Process. Educ Behav. 2012;44:360-364. 1991;50:179-211.
- [Background] Wyker BA, Jordan P, Quigley DL. Evaluation of supplemental nutrition assistance program education: application of behavioral theory and survey validation. J Nutr Educ Behav. 2012 Jul-Aug;44(4):360-4. doi: 10.1016/j.jneb.2011.11.004. Epub 2012 Apr 14. PMID 22507258
- [Background] United States Department of Agriculture, Food and Nutrition Service. About FNS. 2017. Available at: https://www.fns.usda.gov/.(Accessed on 23 May 2021).
- [Background] Dannefer R, Abrami A, Rapoport R, Sriphanlop P, Sacks R, Johns M. A Mixed-Methods Evaluation of a SNAP-Ed Farmers' Market-Based Nutrition Education Program. J Nutr Educ Behav. 2015 Nov-Dec;47(6):516-525.e1. doi: 10.1016/j.jneb.2015.08.021. PMID 26566096
- [Background] Rosemond TN, Blake CE, Shapiro CJ, Burke MP, Bernal J, Adams EJ, Frongillo EA. Disrupted Relationships, Chaos, and Altered Family Meals in Food-Insecure Households: Experiences of Caregivers and Children. J Acad Nutr Diet. 2019 Oct;119(10):1644-1652. doi: 10.1016/j.jand.2019.05.005. Epub 2019 Jul 10. PMID 31302036
- [Background] Burke MP, Martini LH, Blake CE, Younginer NA, Draper CL, Bell BA, Liese AD, Jones SJ. Stretching Food and Being Creative: Caregiver Responses to Child Food Insecurity. J Nutr Educ Behav. 2017 Apr;49(4):296-303.e1. doi: 10.1016/j.jneb.2016.11.010. Epub 2017 Jan 7. PMID 28073623
- [Background] Jomaa L, Na M, Eagleton SG, Diab-El-Harake M, Savage JS. Caregiver's Self-Confidence in Food Resource Management Is Associated with Lower Risk of Household Food Insecurity among SNAP-Ed-Eligible Head Start Families. Nutrients. 2020 Jul 31;12(8):2304. doi: 10.3390/nu12082304. PMID 32751930
- [Background] Gray VB, Hardman AM, Byrd SH. Qualitative Evaluation of Drivers of Eating Decisions among SNAP Participants in Mississippi. J Nutr Educ Behav. 2020 Aug;52(8):775-787. doi: 10.1016/j.jneb.2020.04.006. Epub 2020 Jun 2. PMID 32507480
- [Background] Burke MP, Jones SJ, Frongillo EA, Blake CE, Fram MS. Parenting styles are associated with overall child dietary quality within low-income and food-insecure households. Public Health Nutr. 2019 Oct;22(15):2835-2843. doi: 10.1017/S1368980019001332. Epub 2019 Jun 17. PMID 31203828
- [Background] Brown R, Ogden J. Children's eating attitudes and behaviour: a study of the modelling and control theories of parental influence. Health Educ Res. 2004 Jun;19(3):261-71. doi: 10.1093/her/cyg040. PMID 15140846
- [Background] Callender C, Velazquez D, Adera M, Dave JM, Olvera N, Chen TA, Alford S, Thompson D. How Minority Parents Could Help Children Develop Healthy Eating Behaviors: Parent and Child Perspectives. Nutrients. 2020 Dec 18;12(12):3879. doi: 10.3390/nu12123879. PMID 33353032
- [Background] U.S. Department of Agriculture, Food Research Initiative Competitive Grants Program. Foundational and Applied Science Program Fiscal Years 2021 and 2022 Request for Applications. Available at: https://nifa.usda.gov/sites/default/files/rfa/FY-2021-2022-AFRI-Foundational-and-Applied-Science-RFA-Final-07172020.pdf (Accessed on 23 May 2021).
- [Background] United States Department of Agriculture, National Agricultural Library. Dietary Reference Intakes (DRI) Reports. Available at: https://www.nal.usda.gov/fnic/dietary-reference-intakes (Accessed on 23 May 2021).
- [Background] Hopkins LC, Tiba S, Westrick M, Gunther C. The Diet Quality of a Sample of Predominantly Racial Minority Children From Low-Income Households Is Lower During the Summer vs School Year: Results From the Project Summer Weight and Environmental Assessment Trial Substudy. J Acad Nutr Diet. 2021 Jan;121(1):112-120. doi: 10.1016/j.jand.2020.06.013. Epub 2020 Aug 14. PMID 32800759
- [Background] National Cancer Institute Division of Cancer Control and Population Sciences. Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool. Epidemiology and Genomics Research Program. Available at: https://epi.grants.cancer.gov/asa24/. (Accessed on 24 May 2021).
- [Background] Kong A, Buscemi J, Stolley MR, Schiffer LA, Kim Y, Braunschweig CL, Gomez-Perez SL, Blumstein LB, Van Horn L, Dyer AR, Fitzgibbon ML. Hip-Hop to Health Jr. Randomized Effectiveness Trial: 1-Year Follow-up Results. Am J Prev Med. 2016 Feb;50(2):136-44. doi: 10.1016/j.amepre.2015.07.008. Epub 2015 Sep 16. PMID 26385162
- [Background] Dave JM, Liu Y, Chen TA, Thompson DI, Cullen KW. Does the Kids Cafe Program's Nutrition Education Improve Children's Dietary Intake? A Pilot Evaluation Study. J Nutr Educ Behav. 2018 Mar;50(3):275-282.e1. doi: 10.1016/j.jneb.2017.11.003. Epub 2018 Feb 1. PMID 29395880
- [Background] Dodd KW, Guenther PM, Freedman LS, Subar AF, Kipnis V, Midthune D, Tooze JA, Krebs-Smith SM. Statistical methods for estimating usual intake of nutrients and foods: a review of the theory. J Am Diet Assoc. 2006 Oct;106(10):1640-50. doi: 10.1016/j.jada.2006.07.011. PMID 17000197
- [Background] Kirkpatrick SI, Guenther PM, Douglass D, Zimmerman T, Kahle LL, Atoloye A, Marcinow M, Savoie-Roskos MR, Dodd KW, Durward C. The Provision of Assistance Does Not Substantially Impact the Accuracy of 24-Hour Dietary Recalls Completed Using the Automated Self-Administered 24-H Dietary Assessment Tool among Women with Low Incomes. J Nutr. 2019 Jan 1;149(1):114-122. doi: 10.1093/jn/nxy207. PMID 30602015
- [Background] United States Department of Agriculture, Agricultural Research Service, Food Surveys Research Group. Food and Nutrient Database for Dietary Studies. Available at: https://www.ars.usda.gov/northeast-area/beltsville-md-bhnrc/beltsville-human-nutrition-research-center/food-surveys-research-group/docs/fndds/ (Accessed on 24 May 2021).
- [Background] United States Department of Agriculture, Agricultural Research Service, Food Surveys Research Group. Food Patterns Equivalents Database. Available at: https://www.ars.usda.gov/northeast-area/beltsville-md-bhnrc/beltsville-human-nutrition-research-center/food-surveys-research-group/docs/fped-overview/ (Accessed on 24 May 2021).
- [Background] Sallis JF, Pinski RB, Grossman RM, Patterson TL, Nader PR. The development of self-efficacy scales for health related diet and exercise behaviors. Health education research 1988;3(3):283-92.
- [Background] Savoie MR, Mispireta M, Rankin LL, Neill K, LeBlanc H, Christofferson D. Intention to change nutrition-related behaviors in adult participants of a Supplemental Nutrition Assistance Program-Education. J Nutr Educ Behav. 2015 Jan-Feb;47(1):81-5. doi: 10.1016/j.jneb.2014.08.009. Epub 2014 Sep 27. PMID 25270972